CLINICAL TRIAL: NCT04312581
Title: Effect of Extracorporeal Shock Wave Therapy on Wrist and Hand Functions in Spastic Chronic Stroke Patients :Randomized Controlled Study
Brief Title: Extracorporeal Shock Wave Therapy on Wrist and Hand Functions in Spastic Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, samar abd alhamed tabra, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2020-03-12; First posted 2020-03-18 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Spasticity; Shock Wave
Keywords: shock wave
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (shock wave) (Experimental): Extracorporeal shock wave therapy
  Interventions: Device: Extracorporeal shock wave therapy
- Second group (conventional rehabilitation) (Active Comparator): conventional rehabilitation
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — 3 sessions of radial- extracorporeal shock wave therapy rESWT one week apart, 2000-3000 impulses at 0.25-0.84 millijoule /mm2with a pressure 2.8 bar and 15 Hz frequency.
  Arms: First group (shock wave)
Other: Conventional rehabilitation — physical & occupational therapy
  Arms: Second group (conventional rehabilitation)

SUMMARY:
40 chronic stroke patients with upper limb spasticity will randomly divided into two groups. First group will receive 3 sessions of radial extracorporeal shock wave therapy (rESWT) with one week apart without cessation of current physical therapy, while the second group will continue to receive conventional rehabilitative program.

Assessment will be done at baseline, 2 weeks after rESWT and 3 months after rESWT using Modified Ashworth Scale, Fugl Meyer Assessment for hand function and wrist control, motricity index for pinch grip and Hmax/ Mmax amplitude ratio of flexor carpi radialis muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stroke with disease duration more than one year will be included in the study with stable modified Ashworth scale for upper limb spasticity ranged from 1+ to 4.

Exclusion Criteria:

* Patients more than 65 years,Patients with double stroke and patients with fixed contractures of wrist & hand ,Patients received anti-spastic measures (botulinum toxins, nerve block) within 6 months,Also patients with contraindication to extra-corporeal shock wave therapy i.e. malignancy at treatment area, coagulopathies, active infection (viral or TB), o bleeding wounds, and patients with pacemakers will be excluded

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Change from Pre to Post 1 [after 3rd session (after 2 weeks from baseline) ] and Post 2 (3 months follow-up)
  is a valid scoring system for spasticity
Fugl-Meyer Assessment | Change from Pre to Post 1 [after 3rd session (after 2 weeks from baseline) ] and Post 2 (3 months follow-up)
  reliable assessment tool for sensorimotor function of the upper extremity of stroke patients
Motricity Index | Change from Pre to Post 1 [after 3rd session (after 2 weeks from baseline) ] and Post 2 (3 months follow-up)
  used to assess the motor impairment in a patient with stroke, only one item (pinch grip) was tested using a 2.5 cm cube between the thumb and forefinger
  * 19 points are given if able to grip cube but not hold it against gravity
  * 22 points are given if able to hold cube against gravity but not against a weak pull
  * 26 points are given if able to hold the cube against a weak pull but strength is weaker than normal
Hmax / Mmax amplitude ratio | Change from Pre to Post 1 [after 3rd session (after 2 weeks from baseline) ] and Post 2 (3 months follow-up)
  H reflex is an electrically triggered spinal reflex with a fairly constant latency and amplitude on repeated testing.Hmax / Mmax amplitude ratio was obtained from patient's spastic upper limb, flexor carpi radials muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university hospital, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li TY, Chang CY, Chou YC, Chen LC, Chu HY, Chiang SL, Chang ST, Wu YT. Effect of Radial Shock Wave Therapy on Spasticity of the Upper Limb in Patients With Chronic Stroke: A Prospective, Randomized, Single Blind, Controlled Trial. Medicine (Baltimore). 2016 May;95(18):e3544. doi: 10.1097/MD.0000000000003544. PMID 27149465
- See also: Effect of Radial Shock Wave Therapy on Spasticity of the Upper Limb in Patients With Chronic Stroke — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4863782/